CLINICAL TRIAL: NCT04509726
Title: Single-Arm Trial of EBV Specific Cytokine Secreting TCR-T Cells in the Treatment of EBV-Positive Head and Neck Carcinoma Metastatic/Refractory Nasopharyngeal Carcinoma
Brief Title: EBV Specific Cytokine Secreting TCR-T Cells in the Treatment of EBV-Positive Metastatic/Refractory Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: TCRCure Biopharma Ltd. (Industry)
Responsible Party: Principal Investigator, Qingzhu Jia, M.D., Doctor, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XQDC20200801
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBV TCR-T (Experimental)
  Interventions: Drug: EBV-specific TCR-T cell with cytokine auto-secreting element

INTERVENTIONS:
Drug: EBV-specific TCR-T cell with cytokine auto-secreting element — Patients were pre-conditioned with chemotherapy and infused with EBV-specific TCR-T cells with cytokine auto-secreting element

SUMMARY:
Epstein-Barr virus (EBV) infections is known to be a high-risk factor to induce cervical cancers. To date, EBV-related nasopharyngeal carcinoma (NPC) is still a major concern in east Asia, especially in China. Concurrent therapies for NPC have limited response rate and high chance of relapse. However, EBV-induced cancers provided an ideal target for T cell-based immunotherapy due to the non-self origins. Engineered T cells bearing a TCR (TCR-T) that can specifically recognize the presented EBV-epitope become a viable approach to treat this type of cancer. Though engineered T therapies have been well-recognized in hematological cancers, solid cancer treatment has been a major hurdle due to the immune-suppressive tumor microenvironment. Cytokine seemed to represent the ideal candidate for tumor immunotherapy, due to its ability to activate both innate (NK cells) and adaptive immunities. therefore, TCR-T cells armed with a cytokine -secretion element could further enhance the efficacy of TCR-T in solid cancers.

ELIGIBILITY:
Inclusion Criteria:

* Expected to live longer than 12 weeks
* PS 0-2
* Pathology confirmed as EBV positive NPC, either metastatic or recurrent disease
* Creatinine <2.5mg/dl
* ALT/AST is lower than three times ULN.
* No contraindications of leukocyte collection
* Before entering the trial, women must adopt a reliable method of contraception until 30 days after infusion.
* Understand this trial and have signed an informed consent

Exclusion Criteria:

* Patients with symptomatic brain metastasis
* With other uncontrolled malignant tumors.
* Hepatitis B or Hepatitis C activity period, HIV infected patients
* Any other uncontrolled disease that interferes with the trial
* Patients with severe heart and cerebrovascular diseases such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis and cerebral hemorrhage
* Untreated hypertension or hypertensive patients
* A person with a history of mental illness that is difficult to control
* Researchers do not consider it appropriate to participate in this trial
* Patients who have been using immunosuppressive agents for a long time after organ transplants, except for recent or current inhaled corticosteroids
* Subjects who have been pregnant or nursing, or who plan for pregnancy within 2 months of treatment or after the end of treatment
* An illness affects a person who signs a written consent or complies with a study procedure, or who is unwilling or unable to comply with the research requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
The Maximum Tolerated Dose | 8 weeks
  Verify the MTD of TCR-T cells for EBV antigen for treatment. The first nine patients enrolled in this project will be infused in a dose-escalation approach. The first group of patients will receive 5e+6/kg TCR-T cells, the second group will receive 1e+7/kg TCR-T cells, and the third group will receive 5e+7/kg TCR-T cells. The remaining 11 patients will be infused with TCR-Ts in the maximum tolerated dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided